CLINICAL TRIAL: NCT05939531
Title: Development and Feasibility of a Multi-domain Intervention Program for Post-stroke Bone Health (BOUNCE - Bone Health in Older adUlts' iNtervention Post aCute strokE) in Hospital Pengajar Universiti Putra Malaysia (HPUPM)
Brief Title: Multi-domain Intervention Program for Post-stroke Bone Health in Older Adults (BOUNCE)
Acronym: BOUNCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Pengajar Universiti Putra Malaysia (Other)
Collaborators: Ministry of Higher Education, Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JKEUPM-2022-923
Record Dates: First submitted 2023-03-07; First posted 2023-07-11 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Bone Loss; Stroke; Geriatrics
Keywords: Feasibility; Bone Loss; Intervention; Geriatrics; Stroke
MeSH Terms: conditions — Bone Diseases, Metabolic; Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Standard post-stroke care
  Interventions: Behavioral: Standard Care
- Intervention (Experimental): BOUNCE Program
  Interventions: Behavioral: BOUNCE Program

INTERVENTIONS:
Behavioral: BOUNCE Program — Intervention arm: Bone-building exercises will be incorporated into the standard post-stroke exercises, as well as Nutritional intervention consisting of individualized diet plan based on calorie requirement, high-quality protein intake, vitamin D, Calcium and micronutrients with a one-to-one virtual session.
  Arms: Intervention
Behavioral: Standard Care — Standard post-stroke care
  Arms: Standard Care

SUMMARY:
The goal of this feasibility randomized controlled trial is to assess the feasibility and compare the changes in bone mineral density before and after the intervention in post-stroke older adults. The main question[s] it aims to answer are:

* What are the baseline sociodemographic and bone health characteristics of post-stroke older adults in this study?
* Is it feasible to undertake a larger RCT to assess the effectiveness and implementation of BOUNCE program?
* Is there a difference in bone loss between groups?
* Is there a difference in bone turnover markers at baseline and at six months?
* Is there a difference in the incidence of falls and fragility fractures between groups?
* How receptive are post-stroke patients/carers to the use of food/exercise diary?
* What are the perceived motivators and barriers to implementation of BOUNCE program within real clinical settings among healthcare professionals, participants and carers?
* What is the experience of healthcare professionals, participants and carers undergoing BOUNCE program?

Participants will be divided into two groups:

1. Standard care
2. Intervention group (BOUNCE Program) Researchers will compare both groups to see any changes in the bone mineral density and bone turnover markers before and after the intervention.

DETAILED DESCRIPTION:
Stroke causes secondary osteoporosis, falls and fractures. The 2020 Malaysian Stroke Guideline recommends fall and fracture risk assessment in all older stroke patients, but it does not make a firm recommendation on the interventions to address post-stroke bone loss. Stroke increased the risk of fall by 1.5 times compared to the normal population and quadrupled the risk of fracture. Hip fractures will increase the cost for treatment, hospitalization, operation and complicate the rehabilitation process from the stroke itself.

Hence, our study aims to develop and assess the feasibility of a multi-domain intervention (BOUNCE program) for bone health among older adults with acute stroke. A multi-domain non-pharmacological intervention is proposed due to the complex nature of bone loss in older post-stroke patients such as low serum Vitamin D, sarcopenia, frailty, comorbidity, ageing and hemiparesis. Therefore, this study is designed through the 2021 MRC Framework of Developing and Evaluating Complex Intervention and is divided into 3 phases. The first phase is a systematic review to identify evidence on non-pharmacological interventions for post-stroke bone health. Phase 2 is the development and validation of a novel multi-domain intervention protocol for BOUNCE program through an expert consensus development conference. The final phase will be a feasibility trial of BOUNCE program, which is further divided into two components. The first component is a randomized, controlled, single-blinded feasibility trial (RCT) of 6-months intervention (BOUNCE program) versus standard care, which primarily assesses bone loss through bone mineral density and bone turnover markers. The second component is a qualitative analysis through Focused Group Discussions on the feasibility of BOUNCE program among healthcare professionals, patients and carers. The outcome of this study will inform the next step of evaluation, which is a future full RCT to assess the effectiveness and economic studies before it can be implemented widely.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years old and older
* Neurologist diagnosed acute stroke within 90 days
* Has baseline biochemical test upon admission to the ward
* Able to undergo DXA scan
* Modified Rankin Score of 2 to 3
* Able to walk with or without aids

Exclusion Criteria:

* Known underlying malignancy
* Known major depression or severe psychological illness
* Known chronic kidney disease stage 3b (eGFR <45ml/min/1.73m2) or more
* Taken oral glucocorticoids therapy for at least three months
* Presence of cognitive impairment (ECAQ <7)
* Presence of coronary artery syndrome or congestive cardiac failure
* Presence of an uncontrolled respiratory condition
* Underlying malabsorption syndrome
* Underlying conditions other than stroke that impairs mobility (eg Severe Osteoarthritis, Parkinson's Disease, Multiple sclerosis)
* Known osteoporosis or fragility fracture
* Serum phosphate or calcium abnormalities
* Discharge to a nursing home or rehabilitation centre
* Already a participant in another trial/study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Areal Bone Mineral Density (BMD) at the Neck of Femur as measured by Hologic Dual X-ray Absorptiometry in g/cm2 | At baseline and month-6
  To examine the difference in Areal BMD change pre and post-intervention between groups

SECONDARY OUTCOMES:
Recruitment uptake | Throughout study period of average 1 year
  Number of participants randomized among screened
Change in the level Bone Turnover Markers (BTM) as assessed by C-Telopeptide-Cross-Linked Type I Collagen (CTx) in ng/ml and Procollagen Type I N-Terminal Propeptide (PINP) in ng/ml | At baseline and month-6
  To examine the difference of BTM change pre and post-intervention between groups
Retention | Assessment at month-4 and month-6
  Number of participants followed-up among randomized
Treatment adherence | Assessment at month-4 and month-6
  Number of participants who adhere to the nutritional and exercise interventions in each group
Acceptability | Assessment at month-4 and month-6
  Qualitative study using semi-structured interviews (3 Focus group discussions consist of 10 participants, 10 healthcare professionals and 10 carers) on the motivators, barriers and experience of the intervention
Side-effects | Assessment at month-4 and month-6
  Qualitative study using a semi-structured interview on any side effects of the intervention
Falls | Assessment at month-4 and month-6
  Number of participants experiencing falls during the study period as assessed by Falls Diary
Fracture | Assessment at month-4 and month-6
  Number of participants experiencing bone fragility fracture during the study period as assessed by x-ray evidence

CONTACTS AND LOCATIONS:
Overall Officials: Sazlina Shariff-Ghazali, PhD, Study Chair — Universiti Putra Malaysia
Locations (1):
- Hospital Sultan Abdul Aziz Shah, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No